CLINICAL TRIAL: NCT04071093
Title: Trial Clínico. Utilidad Del Telemonitoreo en Pacientes Con IC Como Medio de Apoyo Para la autogestión de la Enfermedad
Brief Title: Home Telemonitoring System for Patients With Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Nacional de Tucuman (Other)
Responsible Party: Principal Investigator, Lucía María Yanicelli, PhD in Exact Sciences and Engineering, Universidad Nacional de Tucuman
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 94
Record Dates: First submitted 2019-08-22; First posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telemonitoring (Other)
  Interventions: Other: Home Telemonitoring System (HTS)
- Usual Care (No Intervention)

INTERVENTIONS:
Other: Home Telemonitoring System (HTS) — The HTS consists of an App that daily collects measurements of weight, blood pressure, heart rate and symptoms (checklist of symptoms questions). The HTS processes the data and generates and sends an alert to the physicians if a risk situation occurs (measurements are outside of normal ranges). The App has also an educational functionality that allows learning about lifestyle, self-care and healthy habits for HF patients. For this purpose, the application: a) has a section that answers frequent questions, b) has a question and answer game about HF, and c) sends educational messages to the patients every day.
  Arms: Telemonitoring

SUMMARY:
This randomized controlled trial compares a home telemonitoring system (HTS) versus usual care during a 90 days follow-up of Heart Failure (HF) ambulatory patients, in order to evaluate if the use of the HTS improves self-care and treatment adherence. The study was reviewed and approved by the Methodological Committee and by the Research Ethics Committee from the Provincial Health System, according to the Declaration of Helsinki. Written informed consent was obtained before randomization.

ELIGIBILITY:
Inclusion Criteria:

* were over 18 years with a primary diagnosis of HF,
* had been hospitalized at least once time as a consequence of a HF decompensation,
* had a Smartphone,
* had access to WiFi,
* had access to a weight scale and to a blood-pressure monitor

Exclusion Criteria:

* illiterate patients,
* had learning difficulties,
* had a cognitive impairment sufficient to interfere with the use of the telemonitoring system, or had a severe depression that could interfere with their quality of life perception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Changes in self-care | 3-month
  Changes in self-care at baseline and end line of the follow-up using the European Heart Self-care Behavior Questionnaire
Changes in treatment adherence | 3-month
  Changes in treatment adherence at baseline and end line of the follow-up using the Morisky Modified Scale

SECONDARY OUTCOMES:
Rate of Rehospitalizations | 3-month
  Rehospitalizations rate during follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Lucia M Yanicelli, PhD, Principal Investigator — Universidad Nacional de Tucumán
Locations (1):
- Zenón Santillán Health Center Hospital, San Miguel de Tucumán, Tucumán Province, Argentina

REFERENCES:
- [Derived] Yanicelli LM, Goy CB, Gonzalez VDC, Palacios GN, Martinez EC, Herrera MC. Non-invasive home telemonitoring system for heart failure patients: A randomized clinical trial. J Telemed Telecare. 2021 Oct;27(9):553-561. doi: 10.1177/1357633X19899261. Epub 2020 Jan 23. PMID 31973633